CLINICAL TRIAL: NCT06559046
Title: A CT-BASED Deep Learning Model for Predicting WHO/ISUP Pathological Grades of Clear Cell Renal Cell Carcinoma (ccRCC) :A Multicenter Cohort Study
Status: Completed | Type: Observational
Sponsor: Ting Huang (Other)
Responsible Party: Sponsor-Investigator, Ting Huang, Principal Investigator, Zhejiang University
Organization: Zhejiang University (Other)
Other Study IDs: 2024107
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Tumor Grading; Deep Learning; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High grade
- Low grade

SUMMARY:
This study aims to establish an effective deep learning model to extract relevant information about renal tumors and kidneys from computed tomography (CT) images and predict the pathological grades of clear cell renal cell carcinoma (ccRCC).

Retrospective data were collected from 483 ccRCC patients across three medical centers. Arterial phase and portal venous phase CT images from the dataset were segmented for renal tumors and kidneys. Three convolutional neural networks (CNNs) were employed to extract features from the regions of interest (ROI) in the CT images across multiple dimensions including 3D, 2.5D, and 2D. Least absolute shrinkage and selection (LASSO) regression was used for feature selection. The models were evaluated using receiver operating characteristic (ROC) curves and decision curve analysis (DCA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a single kidney tumor have complete imaging and clinical data
* Contrast-enhanced CT scan within 30 days before surgery
* No treatment was performed before CT examination

Exclusion Criteria:

* Patients with tumor recurrence
* Obvious artifacts on CT images
* The tumor is cystic
* Multiple cysts on the affected kidney affect the delineation of renal parenchyma

Ages: 30 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study recruited three cohorts of patients with pathologically diagnosed ccRCC, including a total of 483 patients who underwent nephrectomy or partial nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
predict the pathological grades of clear cell renal cell carcinoma (ccRCC) | 2019-2024
  AUC curve
predict the pathological grades of clear cell renal cell carcinoma (ccRCC) | 2019-2024
  DCA curve

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Affiliated Jinhua Hospital, Zhejiang University School of Medicine, Jinhua,Zhejiang, China, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No